CLINICAL TRIAL: NCT02888860
Title: Analysis of TLRs and Lectin Gene Polymorphisms. Impact on Yeast Colonization in Hospitalized Patients and on Adaptive Response Against Yeast Glycans
Brief Title: Innate Immunity Gene Polymorphisms and Yeast Colonization
Acronym: Candigene
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2011_33; 2011_33 (Other Grant/Funding Number: French Ministry of Health PHRC national 2011); 2012-A00485-38 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2014-02-28; First posted 2016-09-05 (Estimated); Last update posted 2022-11-04 (Actual); Status verified 2020-08

CONDITIONS: Critical Illness
Keywords: genetic susceptibility; candida infection; colonization
MeSH Terms: conditions — Critical Illness; Genetic Predisposition to Disease; Candidiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Biospecimen Retention: Samples With DNA — whole blood, serum, yeast strains, PBMCs
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Group 1: Patients with candidemia
- Group 2: Patients without colonization during follow up
- Group 3: Patients without colonization at admission, with subsequent colonization during hospitalization
- Group: Patients colonized at admission, and during the whole hospitalization
- Group 5: Patients who develop colonization during hospitalization and become negative at discharge

SUMMARY:
It is proposed to carry out the study in three medical or surgical intensive care units (ICU) in the CHRU, Lille, and the CHU, Besançon. In all patients admitted to these ICU (see Figure 2), a corrected index of colonisation (CIC) will be determined and blood samples will be taken for genotyping of the lectins MBL, Dectin-1 and Galectin-3 and for serology. Over the duration of hospitalisation (on average 28 days) and weekly, fungal colonisation will be assessed in all patients (according to the CIC), and antibodies to yeast glycans will be determined by a simultaneous multiparametric analysis involving several families of natural or synthetic antigens, and the detection of circulating antigens (mannan and β-1,3 glucan).

DETAILED DESCRIPTION:
Determination of the CIC:

The CIC will be determined on admission and then once a week during hospitalisation. This will be carried out on a fixed day for all patients; we will avoid determining the CIC any closer than 2 days apart. It is not planned in this study to modify the therapeutic strategy of the ICU services. The strains isolated will be stored in glycerol solution at -80°C. The specimens for genetic and serological analysis will be stored centrally in a local mycology laboratory.

Genotyping of lectin genes and TLRs:

Two tubes containing 6 ml of blood in EDTA will be taken from each patient for extraction of DNA

Serological study, detection of antibodies to yeast glycans:

10 ml of whole blood will be taken from each patient on the day of inclusion and over the duration of hospitalisation (maximum total quantity of 40 ml). This will be done on a fixed day for all patients; we will avoid sampling any closer than 2 days apart.

Functional tests on peripheral blood mononuclear cells (PBMCs) Taking into account the fact that the results of genotyping will not be available in real time and the need to work with freshly collected cells, a group size of 50 patients in group 2 (negative CIC over the duration of hospitalisation) and 50 patients in group 3 (negative CIC at admission but positive at hospital discharge) will be analysed.

Stimulation tests will be carried out in the presence of whole yeasts or yeast extracts on sub-populations of cells isolated from 20 ml of peripheral blood in EDTA.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, ≥18 years of age, admitted to medical or surgical ICU for a duration of >48 h, irrespective of their colonisation status.

Exclusion Criteria:

* -Patient (or their representative) who refuses to participate in the study or to undergo the procedures required for the investigations (mycological sampling in order to determine the CIC, blood sampling for genotyping of DNA and for serology)
* Previous antifungal treatment (in the 15 days preceding admission to the ICU).
* A CIC value based on an insufficient number of sampled sites (<6).
* Neutropenic patients
* Patients who are receiving immunosuppressants (transplanted, grafted...)
* Patients who do not have universal cover or Social Security cover

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients
Sampling Method: Non-Probability Sample
Enrollment: 2200 (Actual)
Dates: Start 2013-01-03 (Actual); Primary Completion 2021-01-03 (Actual); Study Completion 2021-01-03 (Actual)

PRIMARY OUTCOMES:
Frequency of polymorphisms | From date of inclusion until the last day hospital stay (at once a week)
  the frequency is measured for the association between the presence of a polymorphism and colonization by Candida sp.
  frequency of polymorphisms at least one lectin gene or TLRs between some colonized patients (G5) and the non-colonized patients (G2).

SECONDARY OUTCOMES:
Genotyping of lectin genes and toll-like-receptors (TLRs) | From date of inclusion until the last day hospital stay (at once a week)
  The analysis relates to genetic factors already described for lectins and will also include variants of genes involved in innate immunity host-microorganism interactions such as TLRs
Colonization index | at admission and weekly for at least two weeks after.
  This index is calculated for each patient at the entrance of the service and then once a week until discharge (at least two weeks after admission). This index is the ratio between the number of body sites colonized heavily on the number of body sites explored when at least one colony of Candida spp. was observed.
  The determination of Candida colonization index requires the implementation of several samples from different body sites. The sampled anatomical sites concern
  1. mouth (oropharyngeal swab)
  2. stomach (gastric aspiration)
  3. trachea (tracheal suctioning)
  4. urine
  5. rectum (rectal swab or stool).
Functional tests on peripheral blood mononuclear cells (PBMC) | at admission and weekly for at least two weeks after.
  Functional tests on peripheral blood mononuclear cells (PBMC) obtained from mutated patients for given Innate-immunity genes will be carried out through stimulation tests in the presence of whole yeast or derived-molecules on isolated cell subpopulations.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Mathieu, Prof, Principal Investigator — CHRU de Lille
Locations (6):
- France (6):
  - CHRU de Lille, Lille, Nord
  - Centre hospitalier, Arras
  - Centre hosptialier, Boulogne-sur-Mer
  - CH Schaffner, Lens
  - Hôpital Saint-Philibert, Lomme
  - CH Victor Provo, Roubaix